CLINICAL TRIAL: NCT01158898
Title: A Double-Blind,Randomized, Placebo-controlled, 3-Way Cross Over Study to Evaluate the Efficacy and Safety of 14 Days TPI ASM8 in Subjects With Asthma
Brief Title: Efficacy of TPI ASM8 During a 14-Day Allergen Challenge
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Syntara (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TPI ASM8-207
Record Dates: First submitted 2010-06-17; First posted 2010-07-08 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Asthma
Keywords: Mild to moderate asthma; Allergen inhalation challenge
MeSH Terms: conditions — Asthma | interventions — TPI ASM8

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- TPI ASM8 low dose (Active Comparator)
  Interventions: Drug: TPI ASM8
- TPI ASM8 high dose (Active Comparator)
  Interventions: Drug: TPI ASM8
- Placebo (Placebo Comparator)
  Interventions: Drug: TPI ASM8

INTERVENTIONS:
Drug: TPI ASM8 — ASM8 4mg/mL (low dose) daily for 14 days by inhalation
  Arms: TPI ASM8 low dose
Drug: TPI ASM8 — ASM8 4mg/mL (high dose) daily for 14 days by inhalation
  Arms: TPI ASM8 high dose
Drug: TPI ASM8 — Placebo PBS solution daily for 14 days by inhalation
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, 3-way crossover trial to evaluate the efficacy and safety of two different doses of inhaled TPI ASM8 administered daily for 14 days for the treatment of allergic asthma and allergen-induced asthma.

DETAILED DESCRIPTION:
Two doses of TPI ASM8 will be compared to placebo and look at the effect on asthmatic responses after an allergen challenge during a 3-way cross over design. Sputum inflammation , mRNA gene expression on target receptors, ECP , biomarkers of mast cells activation et PK profile will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Mild asthma, male and female aged 18-55 y.old
* Steroid-naive, non-smoker
* Dual responders

Exclusion Criteria:

* Any chronic disease(unstable)
* Immunosuppressed, recent or ongoing steroid intake
* Methacholine PC 20 > 16 mg/mL

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Compare the AUC of the late asthmatic response (LAR) between treatments and placebo | Day 14 (Between 3-7 hr post-AIC)
  The area under the curve fo the late asthmatic response(% fall in FEV1)(between 3-7 hrs post allergen challenge) will be compared between the 2 doses of TPI ASM8 and the placebo

SECONDARY OUTCOMES:
Compare the early and late asthmatic responses between active treatments and placebo after 14 days treatment | Day 14
  Compare the % fall in FEV1 during the EAR and the LAR post-allergen challenge on Day 14.
Compare the Methacholine Hyperresponsiveness (PC20) between treatment pre and post allergen challenge | Day 13 and Day 15 (Pre & post AIC)
  We will compare the PC20( provocative concentration of methacholine) that cause a 20% fall in FEV1
Effect of ASM8 on mast cells (as measured by specific biomarkers) | Day 14 (pre, post and and peri-AIC)
  The leukotriene E4 and 9-11B PGF2 wil be measured in urine and plasma to determine the level of mast cells activation following the allergen challenge
Sputum inflammation indicators (Eos, neutrophils, etc.) | Day 14 and Day 15
  We will measure the levels of total cell counts and the differential to evaluate the degree of inflammation between treatments and placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Paul O'Byrne, MD, Study Chair — McMaster University; Rene Pageau, M.Sc Pharm, Study Director — Pharmaxis Ltd; Louis-Philippe Boulet, MD, Principal Investigator — Hopital Laval, Quebec; Richard Leigh, MD, Principal Investigator — University of Calgary; Gail M Gauveau, PhD, Principal Investigator — McMaster University; Mark Fitzgerald, MD, Principal Investigator — Vancouver Coastal Health Research Institute
Locations (4):
- Canada (4):
  - Health Research Innovation Centre, Calgary, Alberta
  - Vancouver Coastal Health Research Institute, Vancouver, British Columbia
  - McMaster University, Hamilton, Ontario
  - Laval Centre de Pneumologie Chest Division, Québec, Quebec